CLINICAL TRIAL: NCT03913988
Title: Comparative Effectiveness of Three Lucid Dreaming and Sleep Hygiene Techniques to Reduce Stress in Graduate Students on Clinical Internship
Brief Title: Comparative Effectiveness of Three Lucid Dreaming and Sleep Hygiene Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS3098
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Anxiety
Keywords: Dreaming; Sleep; Dream
MeSH Terms: conditions — Anxiety Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Three group, randomized, controlled design
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LUCID DREAMING, STRESS REDUCTION, SLEEP HYGIENE (Active Comparator): This group will meet for 6 online sessions, every other week, over the 12-week study. Each online session will run for 1 hour. Each of the 6 sessions will consist of the following:
  * Psychoeducation regarding lucid dreaming, stress reduction, and sleep hygiene
  * Practice of lucid dreaming induction techniques
  * Guided visualization
  * Opportunity for participants to discuss their experience with lucid dreaming induction techniques, adherence to the lucid dreaming home exercise program and tracking log, using their dream diaries, and adherence to the sleep hygiene program and tracking log.
  Interventions: Behavioral: Lucid Dream; Behavioral: Stress Reduction; Behavioral: Sleep Hygiene Techniques
- LUCID DREAMING, SLEEP HYGIENE (Active Comparator): This group will meet for 6 online sessions, every other week, over the 12-week study. Each online session will run for 1 hour. Each of the 6 sessions will consist of the following:
  * Psychoeducation regarding lucid dreaming and sleep hygiene
  * Practice of lucid dreaming induction techniques
  * Guided visualization
  * Opportunity for participants to discuss their experience with lucid dreaming induction techniques, adherence to the lucid dreaming home exercise program and tracking log, using their dream diaries, and adherence to the sleep hygiene program and tracking log.
  Interventions: Behavioral: Lucid Dream; Behavioral: Sleep Hygiene Techniques
- SLEEP HYGIENE (Active Comparator): This group will meet for 2 online group sessions and 4 email communications. The 2 online group sessions will each last 1 hour and occur in weeks 1 and 12. The 4 email communications will occur in weeks 3, 5, 7, and 9 and consist of individual communication between each participant and the PI or co-investigator. Each email communication will require 10 minutes of participants' time.
  The control group will be asked to engage in Sleep Hygiene techniques in which they adhere to a recommended protocol and record their adherence in a Sleep Hygiene Tracking Log, requiring 5 minutes per day.
  Through the 2 online sessions and the individual email with the investigators, participants will have the opportunity to discuss their experience with adherence to the sleep hygiene program and tracking log. Investigators will help participants trouble shoot problems adhering to the sleep hygiene protocol.
  Interventions: Behavioral: Sleep Hygiene Techniques

INTERVENTIONS:
Behavioral: Lucid Dream — Lucid dream techniques are a set of strategies to induce the ability to obtain conscious awareness during the dream state and include mental suggestions before sleep.
  Arms: LUCID DREAMING, SLEEP HYGIENE; LUCID DREAMING, STRESS REDUCTION, SLEEP HYGIENE
Behavioral: Stress Reduction — Stress reduction techniques are a set of strategies designed to reduce anxiety and include meditation and guided imagery.
  Arms: LUCID DREAMING, STRESS REDUCTION, SLEEP HYGIENE
Behavioral: Sleep Hygiene Techniques — Sleep hygiene is a set of techniques intended to enhance sleep quality and quantity and include maintaining consistent sleep-wake times and avoiding stimulating activities before bed.

SUMMARY:
In this study, the investigators will compare traditional lucid dream induction techniques, stress reduction strategies, and sleep hygiene across three study groups: (1) lucid dream and stress reduction techniques, and sleep hygiene; (2) lucid dream reduction and sleep hygiene; and (3) sleep hygiene. Participants will be first-year occupational therapy students embarking upon their first full-time 3-month clinical internship. Enrolled participants will be randomized to one of the three groups. The intervention will span 12 weeks and allow for participants to learn about and practice lucid dream induction, stress management, and sleep hygiene in bi-monthly online group sessions and through daily home exercises.

DETAILED DESCRIPTION:
A significant impediment to completing academic health care programs is student stress level, which have been reported to be increasing in the last decade. Many students are not prepared for the rigor and intensity of their first clinical internship and experience exacerbations of stress and anxiety at this time. There is evidence that lucid dream induction methods have effectively alleviated stress and anxiety in veterans with post-traumatic stress disorder, and depression in community dwelling adults. Although lucid dream techniques have been used to manage anxiety in some populations, it has never been used to help health care students on clinical internship experiencing heightened stress levels. In this study, the investigators aim to determine whether lucid dream induction techniques combined with stress management and sleep hygiene could effectively help students on their first clinical internship to better manage stress and anxiety. The investigators hope to gain a greater understanding of which of three study conditions can best alleviate stress and anxiety in participants.

ELIGIBILITY:
Inclusion Criteria:

* Current occupational therapy student attending Columbia University and participating in clinical internship

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Week 12
  The Perceived Stress Scale (PSS) is a 10-item, 6-point, self-report Likert scale (0 = no stress, 5 = high stress) that requires 5 minutes to complete. The scale yields a total score ranging from 0 (no stress) to 50 (highest stress) with scores 25+ indicating a possible stress disorder. The PSS measures stress level in the last month and was intended for use by community-dwelling adults.

SECONDARY OUTCOMES:
Lucidity and Consciousness Dream Scale | Week 12
  The Lucidity and Consciousness Dream Scale (LuCiD) is a 28-item, 6-point self-report Likert scale (0 = strongly disagree, 5 = strongly agree) that requires 10 minutes to complete. The scale yields a total score ranging from 0 (no experience of lucid dreaming) to 140 (highest experience of lucid dreaming) with scores 70+ indicating moderate to high lucid dream activity.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, PhD, OTR, FAOTA, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No